CLINICAL TRIAL: NCT02027142
Title: Symptomatic Endometriosis of the Posterior Cul-de-sac is Associated With Impaired Sleep Quality, Excessive Daytime Sleepiness and Insomnia: a Case-control Study.
Brief Title: Sleep Quality, Daytime Sleepiness and Insomnia in Patients With Endometriosis: a Case-control Study.
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Umberto Leone Roberti Maggiore, MD, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Other Study IDs: Sleep and endometriosis.
Record Dates: First submitted 2014-01-02; First posted 2014-01-03 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Endometriosis; Sleep
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Women referred to two academic centres for the diagnosis and treatment of endometriosis.
  Interventions: Other: Pittsburgh Sleep Quality Index.; Other: Epworth sleepiness scale.; Other: Insomnia Severity Index.; Other: The Endometriosis Health Profile.
- Controls: Women referred to our Institutions because of routine gynaecologic consultations.
  Interventions: Other: Pittsburgh Sleep Quality Index.; Other: Epworth sleepiness scale.; Other: Insomnia Severity Index.

INTERVENTIONS:
Other: Pittsburgh Sleep Quality Index. — Pittsburgh Sleep Quality Index is an effective instrument used to measure the quality and patterns of sleep of patients. It allows evaluating "poor" from "good" sleep by assessing seven domains. A total score ≤ 5 indicated good sleep quality while a total score > 5 was indicated poor sleep quality.
Other: Epworth sleepiness scale. — Epworth sleepiness scale is an 8-item questionnaire developed to measure average daytime sleepiness. A total score ≥ 10 indicates excessive daytime sleepiness.
Other: Insomnia Severity Index. — Insomnia Severity Index is a 7-item questionnaire developed to measure insomnia. A total score between 0 and 7 correspond to not clinically significant insomnia, between 8 and 14 to subthreshold insomnia, between 15 and 21 to clinical insomnia (moderate), between 22 and 28 to clinical insomnia (severe).
Other: The Endometriosis Health Profile. — The Endometriosis Health Profile is a patient generated instrument that evaluates disease-specific health-related quality of life in patients with endometriosis. The questionnaire is administrable to all patients with endometriosis and it consists in 30 items divided in 5 domains (pain, control and powerlessness, emotional well-being, social support and self-image). Each scale for each domain is comprised between 0 (indicating the best health status) and 100 (indicating the worst health status).
  Groups: Cases

SUMMARY:
This study included women referred to two academic centres for the diagnosis and treatment of endometriosis (cases) and women referred to our Institutions because of routine gynaecologic consultations (controls). In this age-matched case-control study, the aimdy was to assess quality of sleep, the average daytime sleepiness and insomnia in patients with endometriosis by using three different self-reported questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Reproductive age Surgical and histological diagnosis of rectovaginal endometriosis

Exclusion Criteria:

Suspicion of endometriosis (based on evaluation of symptoms, gynaecological examination and transvaginal ultrasonography) History of infertility Previous diagnosis of endometriosis Gynaecological, intestinal and urological diseases causing abdominal pain (e.g. pelvic congestion syndrome, bladder pain syndrome) Severe underlying comorbidities (cardiovascular, respiratory, renal, hematological, endocrine, hepatic, gastrointestinal, neurological, or psychiatric) Pregnancy at any gestational age Suspicion or diagnosis of oncological pathology Use of gonadotropin releasing hormone analogues (GnRH-a) Restless legs syndrome Shift work Use of antiallergic drugs Narcotics Refusal or inability to sign the informed consent form or complete the study questionnaires

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: In this study were recruited women referred to two academic centres for the diagnosis and treatment of endometriosis (cases) and women referred to our Institutions because of routine gynaecologic consultations (controls).
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Quality of sleep. | Cases were administered and fulfilled the questionnaires at the moment of being scheduled for surgery (3-4 months before the operation). Controls were administered and fulfilled the questionnaires after routine gynaecologic consultation.
  Quality of sleep was assessed by using the Pittsburgh Sleep Quality Index.

SECONDARY OUTCOMES:
Average daytime sleepiness. | Cases were administered and fulfilled the questionnaires at the moment of being scheduled for surgery (3-4 months before the operation). Controls were administered and fulfilled the questionnaires after routine gynaecologic consultation.
  Average daytime sleepiness was assessed by using the Epworth sleepiness scale.
Insomnia. | Cases were administered and fulfilled the questionnaires at the moment of being scheduled for surgery (3-4 months before the operation). Controls were administered and fulfilled the questionnaires after routine gynaecologic consultation.
  Insomnia was assessed by using the Insomnia Severity Index.

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Leone Roberti Maggiore, MD, Principal Investigator — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy; Simone Ferrero, PhD, Study Director — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy; Stefano Salvatore, MD, Principal Investigator — IRRCS San Raffaele Hospital and Vita-Salute San Raffaele University of Milan
Locations (2):
- Italy (2):
  - IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Ligury
  - IRRCS San Raffaele Hospital and Vita-Salute San Raffaele University, Milan, Lombardy